CLINICAL TRIAL: NCT00036959
Title: Phase I Trial and Pharmacokinetic Study of ABT-751, an Orally Bioavailable Tubulin Binding Agent, on a 7 Day and 21 Day Dosing Schedule in Pediatric Patients With Refractory Solid Tumors
Brief Title: ABT-751 in Treating Young Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 020141; 02-C-0141; ABBOTT-M01-357; CDR0000069344; NCT00032266 (obsolete NCT alias)
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Brain and Central Nervous System Tumors; Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Kidney Cancer; Liver Cancer; Neuroblastoma; Ovarian Cancer; Sarcoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: metastatic osteosarcoma; childhood infratentorial ependymoma; recurrent childhood rhabdomyosarcoma; childhood supratentorial ependymoma; childhood craniopharyngioma; disseminated neuroblastoma; recurrent neuroblastoma; recurrent childhood liver cancer; stage IV childhood liver cancer; recurrent Wilms tumor and other childhood kidney tumors; stage IV Wilms tumor; childhood central nervous system germ cell tumor; recurrent osteosarcoma; unspecified childhood solid tumor, protocol specific; childhood germ cell tumor; metastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; childhood high-grade cerebral astrocytoma; childhood oligodendroglioma; childhood choroid plexus tumor; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; recurrent childhood visual pathway and hypothalamic glioma; previously treated childhood rhabdomyosarcoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent childhood ependymoma; childhood teratoma; childhood malignant testicular germ cell tumor; childhood malignant ovarian germ cell tumor; childhood extragonadal germ cell tumor; recurrent childhood malignant germ cell tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Kidney Neoplasms; Liver Neoplasms; Neuroblastoma; Ovarian Neoplasms; Sarcoma; Osteosarcoma; Wilms Tumor; Astrocytoma; Oligodendroglioma; Choroid Plexus Neoplasms; Medulloblastoma; Optic Nerve Glioma; Neuroectodermal Tumors, Primitive, Peripheral; Familial ependymoma; Teratoma; Testicular Neoplasms; Ovarian Germ Cell Cancer | interventions — ABT751

INTERVENTIONS:
Drug: ABT-751

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ABT-751, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase I trial is studying the side effects of ABT-751 in treating young patients with refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and dose-limiting toxic effects of ABT-751 administered daily for 7 days every 21 days or daily for 21 days every 28 days in children with refractory solid tumors.
* Determine the toxicity spectrum of these regimens in these patients.
* Determine the pharmacokinetics of these regimens in these patients.
* Evaluate the pharmacodynamics of this drug by measuring the fraction of tubulin that is polymerized in the peripheral blood mononuclear cells of these patients before and after receiving this drug.

Secondary

* Quantify responses in patients treated with these regimens.
* Assess the effect of this drug on tumor vascularity and tumor blood flow using dynamic enhanced MRI in these patients.

OUTLINE: This is an open-label, multicenter, dose-escalation study of 2 different schedules of ABT-751. Patients are assigned to 1 of 2 dosing schedules.

* Schedule 1 (closed to accrual as of 5/25/2009): Patients receive oral ABT-751 once daily on days 1-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
* Schedule 2 (closed to accrual as of 5/25/2009): Patients receive oral ABT-751 once daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

On each schedule, cohorts of 3-6 patients receive escalating doses of ABT-751 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, up to 9 patients (a minimum of 3 patients age 11 and under and 3 patients age 12 to 18) are treated at the MTD.

PROJECTED ACCRUAL: A maximum of 90 patients will be accrued for this study within 8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor*, including, but not limited to, the following:

  * Rhabdomyosarcoma
  * Other soft tissue sarcomas
  * Ewing's sarcoma family of tumors
  * Osteosarcoma
  * Neuroblastoma
  * Wilms' tumor
  * Hepatic tumors
  * Germ cell tumors
  * Primary brain tumors
  * Brain stem or optic gliomas (histological confirmation may be waived if a biopsy has not been performed) NOTE: *Closed to accrual for all diagnoses except neuroblastoma as of 4/16/05
* Relapsed after or failed to respond to frontline standard therapy and no other standard treatment options (e.g., surgery, radiotherapy, chemotherapy, or any combination of these modalities) exist
* Measurable or evaluable disease* NOTE: *Not required for patients with neuroblastoma
* No CNS tumor with motor or sensory deficits that would obscure the study assessment of sensory neuropathy

PATIENT CHARACTERISTICS:

Age:

* 18 and under

Performance status:

* Lansky 60-100% (age 10 and under)
* Karnofsky 60-100% (age 11 to 18)

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT and AST no greater than 2.5 times ULN (5 times ULN for patients treated after the maximum tolerated dose is determined)
* No clinically significant hepatic dysfunction

Renal:

* Creatinine normal for age OR
* Creatinine clearance at least 60 mL/min
* No clinically significant renal dysfunction

Cardiovascular:

* LVEF normal by echocardiogram

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No allergy to sulfa-containing medications
* No clinically significant unrelated systemic illness (e.g., other organ dysfunction) that would preclude study participation
* No serious infection
* No preexisting grade 2 or greater sensory or motor neuropathy
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 months since prior bone marrow transplantation
* At least 72 hours since prior interleukin-11
* At least 72 hours since prior colony-stimulating factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF]) except epoetin alfa
* No concurrent growth factors (e.g., GM-CSF) except epoetin alfa

  * Concurrent G-CSF allowed if neutropenia lasts longer than 5 days OR if the patient experiences confirmed septicemia associated with neutropenia
* No concurrent immunotherapy
* No concurrent interleukin-11

Chemotherapy:

* See Disease Characteristics
* At least 30 days since prior chemotherapy (42 days for nitrosoureas)
* No other concurrent anticancer chemotherapy

Endocrine therapy:

* Patients with brain tumors:

  * Must be on a stable or tapering dose of corticosteroids for 7 days before baseline scan performed for the purpose of assessing response to study therapy
  * Concurrent corticosteroids allowed for control of symptoms of tumor-associated edema

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* At least 4 months since prior extensive radiotherapy (craniospinal radiotherapy, total body irradiation, or radiotherapy to more than 50% of the pelvis)
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* Recovered from prior therapy
* At least 30 days since prior investigational anticancer therapy
* No other concurrent investigational agents

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2002-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Fox, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Fox E, Maris JM, Cohn SL, Goodspeed W, Goodwin A, Kromplewski M, Medina D, Xiong H, Krivoshik A, Widemann B, Adamson PC, Balis FM. Pharmacokinetics of orally administered ABT-751 in children with neuroblastoma and other solid tumors. Cancer Chemother Pharmacol. 2010 Sep;66(4):737-43. doi: 10.1007/s00280-009-1218-z. Epub 2010 Jan 1. PMID 20044751
- [Result] Fox E, Maris JM, Widemann BC, Goodspeed W, Goodwin A, Kromplewski M, Fouts ME, Medina D, Cohn SL, Krivoshik A, Hagey AE, Adamson PC, Balis FM. A phase I study of ABT-751, an orally bioavailable tubulin inhibitor, administered daily for 21 days every 28 days in pediatric patients with solid tumors. Clin Cancer Res. 2008 Feb 15;14(4):1111-5. doi: 10.1158/1078-0432.CCR-07-4097. PMID 18281544
- [Result] Fox E, Maris JM, Widemann BC, Meek K, Goodwin A, Goodspeed W, Kromplewski M, Fouts ME, Medina D, Cho SY, Cohn SL, Krivoshik A, Hagey AE, Adamson PC, Balis FM. A phase 1 study of ABT-751, an orally bioavailable tubulin inhibitor, administered daily for 7 days every 21 days in pediatric patients with solid tumors. Clin Cancer Res. 2006 Aug 15;12(16):4882-7. doi: 10.1158/1078-0432.CCR-06-0534. PMID 16914576